CLINICAL TRIAL: NCT02934594
Title: Metastatic Spinal Cord Compression (MSCC): Treatment Timing and Survival Rate
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201608007RIND
Record Dates: First submitted 2016-10-11; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Neoplasm Metastasis; Spinal Cord Compression
MeSH Terms: conditions — Neoplasm Metastasis; Spinal Cord Compression

STUDY DESIGN:
Observational Model: Case-Only
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group A: Motor function intact group: received palliative decompression
  Interventions: Other: Palliative Decompression
- Group B1: motor deficit group: received palliative decompression within 48 hours after symptoms occured
  Interventions: Other: Palliative Decompression
- Group B2: motor deficit group: received palliative decompression 48 hours after symptoms occured
  Interventions: Other: Palliative Decompression

INTERVENTIONS:
Other: Palliative Decompression — palliative decompression to MSCC patients: before motor deficit (Group A), within 48 hours after motor deficit (Group B1), 48 hours after motor deficit (Group B2)

SUMMARY:
Patients with metastatic spinal cord compression (MSCC) are treated with different options according to the life expectancy. Survival and surgical outcome can be influenced by surgical timing in MSCC patients treated with palliative decompression.

DETAILED DESCRIPTION:
MSCC patients who underwent palliative decompression after January 2012 in National Taiwan University Hospital (NTUH) were divided into the preoperative motor function intact group (Group A) and motor deficit group (Group B). The motor deficit group was subdivided into operation within 48 hours (Group B1), and after 48 hours (Group B2). All patients underwent palliative decompression and posterior stabilization. Investigators did wide laminectomy for tumor invading the vertebral body, and debulking surgery for tumor destructing the posterior column of the spine. Investigators retrospectively reviewed all patient records, including patient demographics, prognostic factors for survival (Kaplan-Meier survival analysis), neurological outcome (Frankel grade), primary tumor, complications, and relevance of Tomita and Tokuhashi scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic spinal cord compression (MSCC) who underwent palliative decompression in National Taiwan University Hospital after January 1st, 2012.

Exclusion Criteria:

* Patients with metastatic spinal cord compression (MSCC) who underwent palliative decompression before December 31st, 2011, or those who were not treated in National Taiwan University Hospital.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic spinal cord compression (MSCC) who underwent palliative decompression.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
survival rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hua Yang, M.D., Ph.D., Study Chair — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tokuhashi Y, Matsuzaki H, Oda H, Oshima M, Ryu J. A revised scoring system for preoperative evaluation of metastatic spine tumor prognosis. Spine (Phila Pa 1976). 2005 Oct 1;30(19):2186-91. doi: 10.1097/01.brs.0000180401.06919.a5. PMID 16205345
- [Background] Tomita K, Kawahara N, Kobayashi T, Yoshida A, Murakami H, Akamaru T. Surgical strategy for spinal metastases. Spine (Phila Pa 1976). 2001 Feb 1;26(3):298-306. doi: 10.1097/00007632-200102010-00016. PMID 11224867